CLINICAL TRIAL: NCT01274923
Title: The Effect of Low Intensity Shock Wave Therapy on Erectile Dysfunction in Patients Responding to PDE5i's
Brief Title: Double Blind Placebo Controlled Study on the Effect of Extracorporal Shock Wave Therapy on Erectile Dysfunction in PDE5i Responders
Acronym: LI-ESWT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Medispec (Industry)
Responsible Party: Prof Yoram Vardi, Rambam Healthcare Campus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0200-09-rmb europe
Record Dates: First submitted 2011-01-09; First posted 2011-01-12 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-01

CONDITIONS: Erectile Dysfunction
Keywords: Erectile dysfunction; Low Intensity Shock Wave
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- shock wave treatment (Sham Comparator)
  Interventions: Device: "MEDISPEC" treatment probe
- "MEDISPEC" Sham (Sham Comparator): "MEDISPEC" Probe does not deliver energy but creates same noise and sensation of active probe
  Interventions: Device: "MEDISPEC" treatment probe

INTERVENTIONS:
Device: "MEDISPEC" treatment probe — shock wave treatment
  Other Names: Omnispec model ED1000

SUMMARY:
This study aims to evaluate the effect of shockwave therapy on erectile dysfunction on patients responding to PDE5i therapy in a sham controlled randomized double blind manner.

DETAILED DESCRIPTION:
This study aims to evaluate the effect of a 12-session low intensity shockwave therapy protocol for patients with erectile dysfunction. On screening patients will undergo evaluation by thorough medical history and by questionnaires for evaluation of sexual function. A one-month active treatment with PDE5i will be provided followed by re-evaluation using the same questionnaires. Then another one-month period without PDE5i medication (washout period ) will be done and finally on the following visit evaluation will include the same questionnaires and if fit for inclusion- additional objective evaluation of endothelial function using the Flow mediated dilatation technique and penile blood flow measurement by doppler ultrasound of the Penis will be performed. At the end of this screening pahse the first shock wave session will be performed. Altogether 12 treatment sessions will be performed - 6 treatments twice a week followed by a 3 week no-treatment interval and again 6 treatments twice a week. Follow-up which will include the same evaluation as in the first treatment visit will be performed one month after end of treatment

ELIGIBILITY:
Inclusion Criteria:

* ED of more than 6 months
* Rigidity score ≥ 3 under PDE5i therapy
* SHIM ≤21 under PDE5i therapy
* Non- hormonal, neurological or psychological pathology
* Stable heterosexual relationship for more than 3 months

Exclusion Criteria:

* Prior prostatectomy surgery
* Any unstable medical, psychiatric, spinal cord injury and penile anatomical abnormalities
* Clinically significant chronic hematological disease
* Anti-androgens, oral or injectable androgens
* Radiotherapy in pelvic region

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile function- Erectile Function Domain | At screening and 17 weeks later at last visit
  An increase in score of 5points and above will be considered success.

SECONDARY OUTCOMES:
Rigidity scale | At screening and 17 weeks later at last visit
  A change from 1,2 to a result of 3 or 4 of the rigidity scale points will be considered success
Flow Mediated Dilatation Technique | At screening and 17 weeks later at last visit
  A specialized sphygmomanometer cuff located at the penile base, is inflated to 50 mm Hg for 5min to induce a venous filling. A mercury strain gauge is placed at least 1-2 cm above the penile cuff. Baseline penile blood flow is obtained. Postischemic penile blood flow is then recorded immediately after the deflation, until a return to baseline flow is observed. An increase in blood flow above 30% will be considered success.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Haifa District, Israel